CLINICAL TRIAL: NCT00227071
Title: The Effect of Water Verses Land Exercise to Decrease Fall Risk in Older Women With Osteoporosis
Brief Title: Aquatic Verses Land Exercise to Decrease Fall Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Saskatchewan Health Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: BMC 1999-65
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2006-01-04 (Estimated); Status verified 2005-09

CONDITIONS: Osteoporosis
Keywords: accidental falls; osteoporosis; risk factors
MeSH Terms: conditions — Osteoporosis | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
Compare the effect of aquatic,land and no exercise on fall risk factors in women diagnosed with osteoporosis

DETAILED DESCRIPTION:
Background and Purpose: Fall prevention through exercise is an ongoing goal of researchers and clinicians. This study compared the effects of aquatic exercise (AE), land exercise (LE) and no exercise (NE) on fall risk factors. Subjects: Seventy-three women, 60 or older, with osteoporosis (OP). Method: Randomized clinical trial comparing balance, posture, strength, mobility, function, falls, and quality of life. Results: Significant differences (p<0.05) were found for participants' ratings of global change (AE and LE > NE), tandem balance (AE > LE) and function (LE > AE). Joint pain and falls occurred more often during LE. Discussion and Conclusion: Participants experienced significant global improvement with both AE and LE. Less joint pain, reduced falls and improved balance were found in AE, however LE was more effective in improving functional ability at home. Clinicians should consider the individual's specific impairments and risk factors when recommending exercise programs on land or in water.

ELIGIBILITY:
Inclusion Criteria:

* age 60 or older
* diagnosed with osteoporosis
* female

Exclusion Criteria:

* has not been involved in regular exercise in past 2 months
* does not have any medical or neurological condition that would significantly limit activities of daily living, such that involvement in an exercise program would jeopardize safety

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73
Dates: Start 1999-09; Study Completion 2002-06

PRIMARY OUTCOMES:
muscle strength
balance
mobility
function
quality of life

SECONDARY OUTCOMES:
bone status

CONTACTS AND LOCATIONS:
Overall Officials: Cathy M Arnold, Principal Investigator — University of Saskatchewan
Locations (1):
- School of Physical Therapy, Saskatoon, Saskatchewan, Canada